CLINICAL TRIAL: NCT02263014
Title: Treatment Decisions and Breast Cancer: Psychosocial Outcomes
Brief Title: Psychosocial Outcomes and Contralateral Prophylactic Mastectomy (CPM)
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-0752; NCI-2020-07371 (Other: NCI-CTRP Clinical Trials Process Registry)
Record Dates: First submitted 2014-10-08; First posted 2014-10-13 (Estimated); Results first posted 2020-10-05 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Contralateral Prophylactic Mastectomy; Questionnaires; Surveys; Psychosocial
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Contralateral Prophylactic Mastectomy (CPM) Group: Group of women who decide to have contralateral prophylactic mastectomy (CPM) along with scheduled mastectomy. Screening questionnaire completed at baseline. Surgery decision questionnaires completed at surgical consult visit, and at 1, 6, and 12 months after the surgery is completed.
  Interventions: Behavioral: Questionnaires
- No Contralateral Prophylactic Mastectomy (CPM) Group: Group of women who decide not to have contralateral prophylactic mastectomy (CPM) performed during scheduled mastectomy. Screening questionnaire completed at baseline. Surgery decision questionnaires completed at surgical consult visit, and at 1, 6, and 12 months after unilateral mastectomy or breast conserving surgery is completed.
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — Screening questionnaire completed at baseline. Surgery decision questionnaires completed at surgical consult visit, and at 1, 6, 12, and 18 months after the surgery is completed.
  Other Names: Surveys

SUMMARY:
The goal of this research study is to learn more about how different treatment decisions may influence the quality of life in women with breast cancer. Researchers want to use what is learned from this study to help future patients with breast cancer to be more informed when making treatment decisions.

DETAILED DESCRIPTION:
With your verbal permission, you may have been asked to complete a questionnaire about your surgical treatment preferences for breast cancer as part of initial screening for this study. This takes about 5 minutes to complete.

If you agree to participate in this study, during the same visit you will complete a questionnaire about your background, such as your education level, marital status, and family history of cancer. This should take about 3 minutes to complete.

You will also be asked to complete a questionnaire about your surgery decisions and your feelings about those decisions at the following times: around the time you enroll in study before your surgery, and again about 1, 6, and 12 months after the surgery is completed. This questionnaire should take about 30-40 minutes to complete each time. You may complete this questionnaire at the clinic or you may complete it at home. If you chose to complete the questionnaire at home, you will be given a postage-paid envelope to mail it back to the study staff.

Length of Study:

After you complete all of the questionnaires, your participation in this study will be over.

This is an investigational study.

A total of up to 345 participants will be enrolled in this study. Up to 245 will take part at MD Anderson and up to 100 will take part at Kelsey-Seybold.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed ductal carcinoma in situ (DCIS) or Stage I-III sporadic unilateral invasive breast cancer
2. Age 18 or older
3. Able to speak, read, and write English.
4. Spouse/Partner: Married or living with patient for a year or more
5. Spouse/Partner: Age 18 or older
6. Spouse/Partner: Able to speak, read, and write English

Exclusion Criteria:

1. Patients with previous breast cancer
2. Prior history of prophylactic mastectomy
3. Known to have a germline gene mutation that predisposes them to an increased risk of breast cancer (e.g., BRCA1, BRCA2), and/or if they are considered at high risk for contralateral breast cancer on the basis of a strong family history of cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients seen at University of Texas MD Anderson Cancer Center and at Kelsey Seybold Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2014-02-24 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2028-04-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Abenaa M. Brewster, MD, MHS, BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Kelsey-Seybold, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Parker PA, Peterson SK, Shen Y, Bedrosian I, Black DM, Thompson AM, Nelson JC, DeSnyder SM, Cook RL, Hunt KK, Volk RJ, Cantor SB, Dong W, Brewster AM. Prospective Study of Psychosocial Outcomes of Having Contralateral Prophylactic Mastectomy Among Women With Nonhereditary Breast Cancer. J Clin Oncol. 2018 Sep 1;36(25):2630-2638. doi: 10.1200/JCO.2018.78.6442. Epub 2018 Jul 25. PMID 30044695
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: February 24, 2014 to December 31, 2015. All recruitment done at The University of Texas MD Anderson and Kelsey Seybold Clinics.
Pre-assignment Details: Of the 345 women enrolled some were excluded from the study, 37 were determined to be ineligible for participation (reasons included BRCA1/2 carrier, no breast surgery performed, no breast surgery at institutions, metastatic disease at diagnosis) and another 56 women did not complete the required baseline (pre-surgery) assessment.
Groups:
- CPM Group: Contralateral prophylactic mastectomy (CPM) along with scheduled mastectomy. Screening questionnaire completed at baseline. Surgery decision questionnaires completed at surgical consult visit, and at 1, 6, and 12 months after surgery.
- No CPM Group: No CPM performed during scheduled mastectomy. Screening questionnaire completed at baseline. Surgery decision questionnaires completed at surgical consult visit, and at 1, 6, and 12 months after unilateral mastectomy or breast conserving surgery.
Period: Overall Study
Arm/Group | CPM Group | No CPM Group
Started | 44 | 208
Completed | 44 | 208
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- CPM Group: CPM along with scheduled mastectomy. Surgery decision questionnaires completed at surgical consult visit, and at 1, 6, and 12 months after the surgery.
- No CPM Group: No CPM performed during scheduled mastectomy. Surgery decision questionnaires completed at surgical consult visit, and at 1, 6, and 12 months after unilateral mastectomy or breast conserving surgery.
- Total: Total of all reporting groups
Arm/Group | CPM Group | No CPM Group | Total
Number analyzed (Participants) | 44 | 208 | 252
Age, Continuous [Mean (Full Range); unit: years] | 50.9 [30 to 75] | 57.4 [25 to 82] | 56 [25 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 208 | 252
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 24 | 38
  Not Hispanic or Latino | 27 | 174 | 201
  Unknown or Not Reported | 3 | 10 | 13
Region of Enrollment [Number; unit: participants]
  United States | 44 | 208 | 252
Stage, Breast Cancer [Number; unit: percentage of participants] — American Joint Committee on Cancer (AJCC) Breast cancer staging: Anatomic stage 0, I, II, III or IV. AJCC staging system provides strategy for grouping participants by prognosis, based on the extent of the tumor (T), the extent of spread to the lymph nodes (N), and the presence of metastasis (M). Once the T, N, and M are determined, they are combined , and an overall stage of 0, I, II, III, IV is assigned from least advanced to more advanced.
  percentage of participants
    0 | 25 | 18.4 | 19.4
    I | 38.6 | 38.2 | 36.5
    II | 27.3 | 38.6 | 36.9
    III | 9.1 | 6.8 | 7.2
Type of Surgery [Number; unit: percentage of participants]
  Bilateral mastectomy | 100 | 0 | 17.5
  Unilateral mastectomy | 0 | 32.7 | 27.0
  Breast conserving surgery | 0 | 67.3 | 55.6

OUTCOME MEASURES:

1. Primary Outcome: Psychosocial Outcomes of CPM Versus no CPM: Cancer Distress Score
Description: Cancer-specific distress was measured with the Impact of Events Scale (IES) to assess 2 common categories of responses to stressful events: intrusion and avoidance. The IES scale consists of 15 items. For the intrusion category (7 items), participants are asked to rate the items on a 4 point scale: 0 (not at all), 1 (rarely), 3 (sometimes), and 5 (often) and the sum is the total score (complete range is 0 to 35). For the avoidance category (8 items), participants are asked to rate the items on a 4 point scale: 0 (not at all), 1 (rarely), 3 (sometimes), and 5 (often) and the sum is the total score (complete range 0 to 40). The total cancer-specific distress score is the sum of the total intrusion score and the total avoidance score (complete range is 0 to 75). The total distress score was averaged for surveys completed at each time point. Higher mean scores indicate greater cancer-specific distress.
Time Frame: Baseline to 12 months post surgery, up to 18 months. Survey administered at 1, 6, 12 months following surgery.
Population: Two participants of the CPM Group (N=44) who had CPM after the date of their primary surgery were excluded from the longitudinal study analysis. *The overall number of patients analyzed may differ from the total number analyzed at each time point since not all surveys were returned at each time point.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- CPM Group: CPM along with scheduled mastectomy. Questionnaires completed at baseline (pre-surgery) and at 1, 6, and 12 months post-surgery.
- No CPM Group: No CPM performed during scheduled mastectomy. Surgery decision questionnaires completed at baseline (pre-surgery), and at 1, 6, and 12 months after unilateral mastectomy or breast conserving surgery.
Arm/Group | CPM Group | No CPM Group
Number analyzed (Participants) | 42 | 208
units on a scale
  Pre-Surgery: number analyzed (Participants) | 42 | 207
  Pre-Surgery | 29.98 (16.77) | 24.62 (16.52)
  1 Month Post-surgery: number analyzed (Participants) | 38 | 189
  1 Month Post-surgery | 21.84 (14.58) | 19.84 (14.8)
  6 Months Post-surgery: number analyzed (Participants) | 40 | 196
  6 Months Post-surgery | 23.43 (14.69) | 18.56 (16.11)
  12 Months Post-surgery: number analyzed (Participants) | 33 | 169
  12 Months Post-surgery | 25.3 (17.26) | 17.01 (14.79)

2. Primary Outcome: Psychosocial Outcomes of CPM Versus no CPM: Satisfaction With Decision
Description: The Satisfaction with Decision Scale (SWD) scale measures women's satisfaction with their surgery decision using the SWD six-item survey with a five-point scale where 1 is "strongly disagree" and 5 is "strongly agree" and the sum is the total score (complete range 6 to 30). The total satisfaction with decision score was averaged for surveys completed at each time point. Higher mean scores indicate greater satisfaction with the treatment decision.
Time Frame: One to 12 months post surgery, up to 18 months. Survey administered at 1, 6, 12 months following surgery.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CPM Group | No CPM Group
Number analyzed (Participants) | 42 | 208
units on a scale
  1 Month assessment: number analyzed (Participants) | 38 | 187
  1 Month assessment | 4.23 (1.08) | 4.27 (0.81)
  6 month assessment: number analyzed (Participants) | 39 | 192
  6 month assessment | 4.18 (1.06) | 4.33 (0.76)
  12 month assessment: number analyzed (Participants) | 32 | 168
  12 month assessment | 4.35 (0.86) | 4.34 (0.75)

ADVERSE EVENTS:
Time Frame: Adverse event data collected up to 12 months following surgery for breast cancer.
Groups:
- CPM Group: CPM along with scheduled mastectomy. Surgery decision questionnaires completed at surgical consult visit, and at 1, 6, and 12 months after surgery.
Arm/Group | CPM Group | No CPM Group
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/208
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/208
Other Adverse Events (participants affected / at risk) | 0/44 | 0/208

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-30): https://cdn.clinicaltrials.gov/large-docs/14/NCT02263014/Prot_SAP_000.pdf